CLINICAL TRIAL: NCT06925945
Title: Comparison of Pain Between Modified Thoracoabdominal Plane Block and Rectus Block Combination and Intraperitoneal Local Infiltration Analgesia
Brief Title: Modified Thoracoabdominal Plane Block and Rectus Block Combination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Hüseyin Demir, MD, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HASEKİ TEZ
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Visual Analogue Scale

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified thoracoabdominal plane block (M-TAPA) and rectus sheath block (Active Comparator): Modified thoracoabdominal plane block (M-TAPA) and rectus sheath block
  Interventions: Procedure: regional anestesia
- local infiltration analgesia (Active Comparator): local infiltration analgesia
  Interventions: Procedure: regional anestesia

INTERVENTIONS:
Procedure: regional anestesia — Modified thoracoabdominal plane block (M-TAPA) and rectus sheath block with local infiltration analgesia

SUMMARY:
The aim of our study was to investigate the effect of the combination of Modified thoracoabdominal plane block (M-TAPA) and rectus sheath block with local infiltration analgesia on postoperative pain scores and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* ASA1-2
* Laparoscopic cholecystectomy cases

Exclusion Criteria:

* Bleeding disorders
* Anticoagulant use
* Patients with previous nerve damage
* Lack of patient consent
* Patients with liver and kidney failure
* Patients allergic to local anesthetics used
* Patients with BMI > 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 4 month
  Pain score measured using a 0-10 scale, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gungor H, Ciftci B, Alver S, Golboyu BE, Ozdenkaya Y, Tulgar S. Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) vs local infiltration for pain management after laparoscopic cholecystectomy surgery: a randomized study. J Anesth. 2023 Apr;37(2):254-260. doi: 10.1007/s00540-022-03158-0. Epub 2022 Dec 28. PMID 36575362
- [Result] Erten E, Kara U, Simsek F, Oztas M, Suzer MA, Kamburoglu H, Eskin MB, Senkal S, Cosar A. Modified thoracoabdominal nerves block through perichondrial approach for laparoscopic cholecystectomy. Rev Assoc Med Bras (1992). 2024 Apr 22;70(3):e20230962. doi: 10.1590/1806-9282.20230962. eCollection 2024. PMID 38655995